CLINICAL TRIAL: NCT05062707
Title: Longitudinal Assessment of Therapy-related Early Ageing in Adolescent and Young Adult (AYA) Cancer Patients
Brief Title: Early Ageing During Therapy in AYA Cancer Patients
Status: Recruiting | Type: Observational
Sponsor: University Medical Center Groningen (Other)
Collaborators: UMCG Kanker Researchfonds (Unknown)
Responsible Party: Sponsor
Other Study IDs: 202100484
Record Dates: First submitted 2021-09-21; First posted 2021-09-30 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Cancer; Leukemia; Hodgkin Lymphoma; Testicular Cancer; Osteosarcoma; Ewing Sarcoma; Breast Cancer; Cervical Cancer
MeSH Terms: conditions — Neoplasms; Leukemia; Hodgkin Disease; Testicular Neoplasms; Osteosarcoma; Sarcoma, Ewing; Breast Neoplasms; Uterine Cervical Neoplasms | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Fasting blood samples (65 ml in total) will be drawn to measure circulating senescence marker P16 (in circulating CD3+ (cluster of differentiation 3+) T-lymphocytes), markers of the SASP (IL-6, IL-8, VEGF (vascular endothelial growth factor) ), biochemical markers for vascular damage (von Willebrand Factor, albuminuria, coagulation markers (i.e.FVIII, fibrinogen, Plasminogen Activator inhibitor -1), high sensitivity C-reactive protein (hs-CRP), NT-proBNP (Brain Natriuretic Peptide), galectin-3, GDF-15 (Growth/Differentiation Factor-15)), and the cardiovascular risk profile (total cholesterol, triglycerides, HDL-cholesterol (high-density lipoprotein), LDL-cholesterol (low density lipoprotein); glucose, insulin, and HbA1c). The investigators will also isolate genomic DNA and RNA from full blood samples to assess SNP (single nucleotide polymorphism)-array and methylation profile as a measure for biological age.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- AYA cancer patients: Patients aged 18-39 years, with a first histological and/or cytological diagnosis of a haematological or solid malignancy, scheduled to start systemic therapy with curative intent.
  Interventions: Procedure: Blood sampling

INTERVENTIONS:
Procedure: Blood sampling — Study measurements will be performed twice and consist of blood withdrawal and physical examination (weight, height, waist-hip ratio, and blood pressure).

SUMMARY:
Longitudinal cohort study; measurements before start of systemic therapy and one year later.

DETAILED DESCRIPTION:
Rationale:

Compared with survivors of childhood cancer, there is sparse knowledge about the long-term morbidity and mortality of adolescent and young adult (AYA) cancer patients, who are diagnosed at age 18-39 and have an 80% chance to survive. Following cancer treatment, many cancer survivors, including those at AYA age, have an increased risk of cardiovascular disease. Early ageing has been described in paediatric and certain adult cancer survivor populations. One of the responsible mechanisms behind biological ageing is cellular senescence, characterized by a stable arrest of the cell cycle which occurs in response to stress and damage. In all organisms the number of senescent cells increases with age and senescence has been associated with age-related diseases, like atherosclerosis and Alzheimer. Early ageing as a result of intensive cancer treatment with systemic therapy and radiation may result in early cardiovascular disease. However, information about senescence, early vascular ageing and related patient and tumour characteristics is missing for AYAs.

Objective:

to determine markers related to early ageing and senescence in AYA cancer patients before and after systemic therapy, in order to assess treatment-related early vascular ageing and associated tumour and patient characteristics.

Study design:

Longitudinal cohort study; measurements before start of systemic therapy and one year later.

Study population:

Patients aged 18-39 years, with a first histological and/or cytological diagnosis of a haematological or solid malignancy, scheduled to start systemic therapy with curative intent.

Main study parameters/endpoints:

Primary endpoint is change in senescence marker P16 between start of systemic therapy and one year later. Secondary endpoints are: changes in senescence-associated secretory phenotype (SASP) and vascular markers; prevalence of classical cardiovascular risk factors (smoking, lipids, body mass index (BMI), glucose); tumour (treatment) and patient (age, sex, pre-existent cardiometabolic status) factors related to the changes in senescence, SASP and cardiovascular risk factors.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: Study measurements will be performed twice and consist of blood withdrawal and physical examination (weight, height, waist-hip ratio, and blood pressure).

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-39 years at cancer diagnosis
* Having a histologically and/or cytologically confirmed cancer diagnosis, including leukemia, (non-)Hodgkin lymphoma, testicular cancer, osteosarcoma, Ewing sarcoma, breast cancer, and cervical cancer.
* Scheduled to start systemic therapy with curative intent. Allowed treatments (concurrent or sequential) are: surgery, radiotherapy, chemotherapy, antibodies.

Exclusion Criteria:

* patients who are not able to understand the patient information letter and informed consent form
* patients who will be treated with immune checkpoint inhibitors or targeted therapy with inhibitors of angiogenesis
* patients who have been treated with systemic therapy or radiotherapy for a previous malignancy (exceptions: in situ carcinoma of the cervix or uterus and adequately treated basal and squamous cell carcinoma of the skin).

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: AYA patients who will start systemic treatment at the Department of Medical Oncology or Haematology of the University Medical Center Groningen are potential study participants. Patients will be informed about the study during a regular visit to the outpatient clinic or during their admission to the nursing ward. From the moment the study starts, the investigators aim to include all consecutive patients during a period of 2 years.
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2022-02-10 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Change in senescence marker P16 | at baseline and 1 year after start systemic therapy
  determine change in senescence marker P16 between start of systemic therapy and one year later.

SECONDARY OUTCOMES:
Changes in SASPs and vascular markers | at baseline and 1 year after start systemic therapy
  Determine changes in SASPs and vascular markers
Prevalence of classical cardiovascular risk factors (smoking, lipids, BMI, glucose) | at baseline and 1 year after start systemic therapy
  Determine prevalence of classical cardiovascular risk factors (lipids, BMI, glucose)
Association between treatment type and change in senescence marker P16 | at baseline and 1 year after start systemic therapy
  Determine association between treatment type and change in senescence marker P16
Association between age and change in senescence marker P16 | at baseline and 1 year after start systemic therapy
  Determine association between age and change in senescence marker P16
Associations between senescence, inflammation, and cardiovascular risk factors | at baseline and 1 year after start systemic therapy
  Determine associations between senescence, inflammation, and cardiovascular risk factors

CONTACTS AND LOCATIONS:
Overall Officials: J. Nuver, MD, PhD, Principal Investigator — University Medical Center Groningen
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands